CLINICAL TRIAL: NCT04752462
Title: Effect of Post-Discharge Telemedicine Motivational Enhancement Intervention in Heart Failure and Obstructive Sleep Apnea on Adherence and Health Outcomes
Brief Title: Motivational Enhancement - Acute Decompensated Heart Failure and OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Cinthya Pena Orbea, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-075
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Decompensated Heart Failure; Obstructive Sleep Apnea; Motivational Enhancement; PAP Adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care with provider (No Intervention): Participant will continue follow up for sleep apnea with provider.
- Telemedicine Intensive Motivational Enhancement (Experimental): Participants will attend a telemedicine motivational enhancement visit to improve PAP adherence along with regular follow up for sleep apnea
  Interventions: Behavioral: Telemedicine Intensive Motivational Enhancement

INTERVENTIONS:
Behavioral: Telemedicine Intensive Motivational Enhancement — Participants will attend a telemedicine motivational enhancement visit to improve PAP adherence along with regular follow up for sleep apnea
  Other Names: TIME
  Arms: Telemedicine Intensive Motivational Enhancement

SUMMARY:
A feasibility randomized controlled trial will be conducted with a 6-month follow up to: Examine the impact of early intensive telemedicine motivational enhancement (TIME) vs standard of care on PAP adherence (n=40/group) and continuity of care at 3 and 6 months post-discharge in patients admitted with ADHF with a new inpatient diagnosis of OSA(REI>5). Assess the effect of early telemedicine integrated with motivational enhancement (TIME) vs standard of care on patient reported outcomes including Functional Outcomes of Sleep questionnaire (FOSQ-10), Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Investigate the impact of early TIME vs standard of care on 6-month hospital readmissions.

DETAILED DESCRIPTION:
As part of our inpatient sleep testing program, high-risk HF patients undergo Type III sleep testing (Nihon Kohden®) set up by sleep laboratory technicians. Our inpatient sleep service also has a clinical nurse who works with patients on CPAP education, set up and assists with post hospital sleep care. If a titration study is needed, it is generally arranged 1-2 weeks post discharge. All inpatient sleep studies are scored by three registered polysomnographic technologists and I review and finalize these studies (current clinical flow as the primary physician leading the inpatient service, which will be augmented for this clinical trial). A research coordinator and I will approach those with REI>5 who meet eligibility per screening in Epic®, to discuss sleep study results, confirm eligibility, invite the patient to participate, and if interested, will obtain written informed consent. Consent: Consent form will explain in a lay person' terminology the nature of all procedures. It will be stressed that participation is voluntary. The research coordinator and the PI will be available to answer questions. All activities will be compliant with local IRB and HIPPA guidelines.

All participants will obtain Auto-CPAP from two manufacturers (Philips Respironics ® or ResMed ®) delivered by the same homecare health before discharge. PAP pressures will be set at 5-15 cmH2O, heated humification, and expiratory pressure relief according to comfort. A modem will be attached to the PAP device to extract adherence data remotely (SD card for those without wireless capability). All patients will receive a standardized 20-minute educational session about PAP therapy before discharge and will be advised to use their device every night during sleep by our clinical nurse. Patients will also be fitted for a mask fitted homecare health. If participants have mask or pressure intolerance issues, they will be a direct provided a phone number to our research coordinator. All baseline questionnaires will be sent via REDcap link to the patient's e-mail or completed in paper form before discharge and during their visit (or paper if electronic not feasible). The coordinator will ensure all questionnaires are completed before discharge and will instruct patients to complete follow-up questionnaires. Patients will be randomized (REDCap algorithm) 1:1 to TIME versus standard of care. Blocks will be of random size blinded to study investigators. Although it will not be feasible to blind the research team and participants to the intervention, the standard of care group will also receive sleep hygiene education so that there is perception of some level of intervention to try to address placebo effect. During follow up visits (2 weeks and 2 months for the TIME group and 2 months standard of care group) with sleep medicine, the first 15 minutes will be focused on OSA and troubleshooting problems for both groups as this is standard clinical care provided at our Sleep Disorders Center. These 15 minutes will be followed by 30 minutes of ME in the intervention group and 10 minutes of sleep hygiene education in the control group. Outcomes will be measured at 3 months and 6 months for both groups. Both groups will receive a booster phone call at 4 months. The intervention group will receive a 30 minutes booster ME session and the control group will receive 10 minutes of sleep hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Admitting ADHF diagnosis
* OSA diagnosis (REI ≥5)
* Treatment-naive and agreeable to PAP therapy
* Agrees to participate.

Exclusion Criteria:

* Prior or current PAP therapy
* Unable to provide informed consent
* Moderately hypoxic (oxygen saturation < 87% on room air or requiring >2L of O2 during overnight sleep study
* Hemodynamically unstable (systolic blood pressure, SBP<90 mmHg, heart rate>120bpm)
* Central predominant apnea (Central Apnea Index > 50% of the Apnea Index) Dementia/cognitive dysfunction
* Unable to participant in video televisits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
PAP Adherence (TIME versus Standard of Care) | 3 Month
  average hourly use per night
PAP Adherence (TIME versus Standard of Care) | 6 Month
  average hourly use per night
Functional Outcomes of Sleep Questionnaire (TIME versus Standard of Care) | 2 Months
  Functional Outcomes of Sleep Questionnaire (FOSQ-10): Subscale scores range from 1-4 (1= extreme difficulty, 2= moderate difficulty, 3= a little difficulty, 4= no difficulty) with total scores ranging from 5-20 with higher scores indicating better functional status.
Kansas City Cardiomyopathy Questionnaire (TIME versus Standard of Care) | 2 Months
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12):: physical limitation, symptom frequency, quality of life, and social limitation. Scores ranges from 5-30, higher KCCQ-12 scores from baseline represent better health status

OTHER OUTCOMES:
Impact of TIME vs Standard of Care on 6-month hospital readmissions | 6 Month
  6-month hospital readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Cinthya Pena Orbea, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] Khayat R, Small R, Rathman L, Krueger S, Gocke B, Clark L, Yamokoski L, Abraham WT. Sleep-disordered breathing in heart failure: identifying and treating an important but often unrecognized comorbidity in heart failure patients. J Card Fail. 2013 Jun;19(6):431-44. doi: 10.1016/j.cardfail.2013.04.005. PMID 23743494
- [Background] Khayat RN, Jarjoura D, Patt B, Yamokoski T, Abraham WT. In-hospital testing for sleep-disordered breathing in hospitalized patients with decompensated heart failure: report of prevalence and patient characteristics. J Card Fail. 2009 Nov;15(9):739-46. doi: 10.1016/j.cardfail.2009.05.005. Epub 2009 Jun 26. PMID 19879459
- [Background] Khattak HK, Hayat F, Pamboukian SV, Hahn HS, Schwartz BP, Stein PK. Obstructive Sleep Apnea in Heart Failure: Review of Prevalence, Treatment with Continuous Positive Airway Pressure, and Prognosis. Tex Heart Inst J. 2018 Jun 1;45(3):151-161. doi: 10.14503/THIJ-15-5678. eCollection 2018 Jun. PMID 30072851
- [Background] Khayat R, Jarjoura D, Porter K, Sow A, Wannemacher J, Dohar R, Pleister A, Abraham WT. Sleep disordered breathing and post-discharge mortality in patients with acute heart failure. Eur Heart J. 2015 Jun 14;36(23):1463-9. doi: 10.1093/eurheartj/ehu522. Epub 2015 Jan 29. PMID 25636743
- [Background] Fox N, Hirsch-Allen AJ, Goodfellow E, Wenner J, Fleetham J, Ryan CF, Kwiatkowska M, Ayas NT. The impact of a telemedicine monitoring system on positive airway pressure adherence in patients with obstructive sleep apnea: a randomized controlled trial. Sleep. 2012 Apr 1;35(4):477-81. doi: 10.5665/sleep.1728. PMID 22467985
- [Background] Isetta V, Leon C, Torres M, Embid C, Roca J, Navajas D, Farre R, Montserrat JM. Telemedicine-based approach for obstructive sleep apnea management: building evidence. Interact J Med Res. 2014 Feb 19;3(1):e6. doi: 10.2196/ijmr.3060. PMID 24554392
- [Background] Hoy CJ, Vennelle M, Kingshott RN, Engleman HM, Douglas NJ. Can intensive support improve continuous positive airway pressure use in patients with the sleep apnea/hypopnea syndrome? Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1096-100. doi: 10.1164/ajrccm.159.4.9808008. PMID 10194151
- [Background] Kitsiou S, Pare G, Jaana M. Effects of home telemonitoring interventions on patients with chronic heart failure: an overview of systematic reviews. J Med Internet Res. 2015 Mar 12;17(3):e63. doi: 10.2196/jmir.4174. PMID 25768664
- [Background] Van Ryswyk E, Anderson CS, Antic NA, Barbe F, Bittencourt L, Freed R, Heeley E, Liu Z, Loffler KA, Lorenzi-Filho G, Luo Y, Margalef MJM, McEvoy RD, Mediano O, Mukherjee S, Ou Q, Woodman R, Zhang X, Chai-Coetzer CL. Predictors of long-term adherence to continuous positive airway pressure in patients with obstructive sleep apnea and cardiovascular disease. Sleep. 2019 Oct 9;42(10):zsz152. doi: 10.1093/sleep/zsz152. PMID 31587046
- [Background] Bakker JP, Weaver TE, Parthasarathy S, Aloia MS. Adherence to CPAP: What Should We Be Aiming For, and How Can We Get There? Chest. 2019 Jun;155(6):1272-1287. doi: 10.1016/j.chest.2019.01.012. Epub 2019 Jan 23. PMID 30684472
- [Background] Bakker JP, Wang R, Weng J, Aloia MS, Toth C, Morrical MG, Gleason KJ, Rueschman M, Dorsey C, Patel SR, Ware JH, Mittleman MA, Redline S. Motivational Enhancement for Increasing Adherence to CPAP: A Randomized Controlled Trial. Chest. 2016 Aug;150(2):337-45. doi: 10.1016/j.chest.2016.03.019. Epub 2016 Mar 24. PMID 27018174
- [Background] Smith CE, Dauz ER, Clements F, Puno FN, Cook D, Doolittle G, Leeds W. Telehealth services to improve nonadherence: A placebo-controlled study. Telemed J E Health. 2006 Jun;12(3):289-96. doi: 10.1089/tmj.2006.12.289. PMID 16796496
- [Background] Rohr R. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Jul 16;361(3):311-2; author reply 312. No abstract available. PMID 19610166
- [Background] Joynt KE, Jha AK. Who has higher readmission rates for heart failure, and why? Implications for efforts to improve care using financial incentives. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):53-9. doi: 10.1161/CIRCOUTCOMES.110.950964. Epub 2010 Dec 14. PMID 21156879
- [Background] Amir O, Ben-Gal T, Weinstein JM, Schliamser J, Burkhoff D, Abbo A, Abraham WT. Evaluation of remote dielectric sensing (ReDS) technology-guided therapy for decreasing heart failure re-hospitalizations. Int J Cardiol. 2017 Aug 1;240:279-284. doi: 10.1016/j.ijcard.2017.02.120. Epub 2017 Mar 3. PMID 28341372
- [Background] Athilingam P, Jenkins BA, Zumpano H, Labrador MA. "Mobile technology to improve heart failure outcomes: A proof of concept paper". Appl Nurs Res. 2018 Feb;39:26-33. doi: 10.1016/j.apnr.2017.10.018. Epub 2017 Oct 19. PMID 29422170
- [Background] McAlister FA, Youngson E, Kaul P, Ezekowitz JA. Early Follow-Up After a Heart Failure Exacerbation: The Importance of Continuity. Circ Heart Fail. 2016 Sep;9(9):e003194. doi: 10.1161/CIRCHEARTFAILURE.116.003194. PMID 27618853
- [Background] MacDonald M, Fang J, Pittman SD, White DP, Malhotra A. The current prevalence of sleep disordered breathing in congestive heart failure patients treated with beta-blockers. J Clin Sleep Med. 2008 Feb 15;4(1):38-42. PMID 18350960
- [Background] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114
- [Background] Wang H, Parker JD, Newton GE, Floras JS, Mak S, Chiu KL, Ruttanaumpawan P, Tomlinson G, Bradley TD. Influence of obstructive sleep apnea on mortality in patients with heart failure. J Am Coll Cardiol. 2007 Apr 17;49(15):1625-1631. doi: 10.1016/j.jacc.2006.12.046. Epub 2007 Apr 2. PMID 17433953
- [Background] Sharma S, Chakraborty A, Chowdhury A, Mukhtar U, Willes L, Quan SF. Adherence to Positive Airway Pressure Therapy in Hospitalized Patients with Decompensated Heart Failure and Sleep-Disordered Breathing. J Clin Sleep Med. 2016 Dec 15;12(12):1615-1621. doi: 10.5664/jcsm.6344. PMID 27568891
- [Background] Kauta SR, Keenan BT, Goldberg L, Schwab RJ. Diagnosis and treatment of sleep disordered breathing in hospitalized cardiac patients: a reduction in 30-day hospital readmission rates. J Clin Sleep Med. 2014 Oct 15;10(10):1051-9. doi: 10.5664/jcsm.4096. PMID 25317084
- [Background] Isetta V, Negrin MA, Monasterio C, Masa JF, Feu N, Alvarez A, Campos-Rodriguez F, Ruiz C, Abad J, Vazquez-Polo FJ, Farre R, Galdeano M, Lloberes P, Embid C, de la Pena M, Puertas J, Dalmases M, Salord N, Corral J, Jurado B, Leon C, Egea C, Munoz A, Parra O, Cambrodi R, Martel-Escobar M, Arque M, Montserrat JM; SPANISH SLEEP NETWORK. A Bayesian cost-effectiveness analysis of a telemedicine-based strategy for the management of sleep apnoea: a multicentre randomised controlled trial. Thorax. 2015 Nov;70(11):1054-61. doi: 10.1136/thoraxjnl-2015-207032. Epub 2015 Aug 26. PMID 26310452
- [Background] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Kirwan BA, Winkler S, Vettorazzi E, Bruch L, Oeff M, Zugck C, Doerr G, Naegele H, Stork S, Butter C, Sechtem U, Angermann C, Gola G, Prondzinsky R, Edelmann F, Spethmann S, Schellong SM, Schulze PC, Bauersachs J, Wellge B, Schoebel C, Tajsic M, Dreger H, Anker SD, Stangl K. Efficacy of telemedical interventional management in patients with heart failure (TIM-HF2): a randomised, controlled, parallel-group, unmasked trial. Lancet. 2018 Sep 22;392(10152):1047-1057. doi: 10.1016/S0140-6736(18)31880-4. Epub 2018 Aug 25. PMID 30153985
- [Background] Aloia MS, Arnedt JT, Stepnowsky C, Hecht J, Borrelli B. Predicting treatment adherence in obstructive sleep apnea using principles of behavior change. J Clin Sleep Med. 2005 Oct 15;1(4):346-53. PMID 17564399
- [Background] Stepnowsky CJ Jr, Marler MR, Ancoli-Israel S. Determinants of nasal CPAP compliance. Sleep Med. 2002 May;3(3):239-47. doi: 10.1016/s1389-9457(01)00162-9. PMID 14592213
- [Background] Olsen S, Smith SS, Oei TP, Douglas J. Motivational interviewing (MINT) improves continuous positive airway pressure (CPAP) acceptance and adherence: a randomized controlled trial. J Consult Clin Psychol. 2012 Feb;80(1):151-63. doi: 10.1037/a0026302. Epub 2011 Nov 21. PMID 22103957
- [Background] Lai AYK, Fong DYT, Lam JCM, Weaver TE, Ip MSM. The efficacy of a brief motivational enhancement education program on CPAP adherence in OSA: a randomized controlled trial. Chest. 2014 Sep;146(3):600-610. doi: 10.1378/chest.13-2228. PMID 24810282
- [Background] Arzt M, Young T, Finn L, Skatrud JB, Ryan CM, Newton GE, Mak S, Parker JD, Floras JS, Bradley TD. Sleepiness and sleep in patients with both systolic heart failure and obstructive sleep apnea. Arch Intern Med. 2006 Sep 18;166(16):1716-22. doi: 10.1001/archinte.166.16.1716. PMID 16983049
- [Background] Kahwash R, Khayat RN. A Practical Approach to the Identification and Management of Sleep-Disordered Breathing in Heart Failure Patients. Sleep Med Clin. 2017 Jun;12(2):205-219. doi: 10.1016/j.jsmc.2017.01.002. Epub 2017 Mar 9. PMID 28477775
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- [Background] Collop NA, Tracy SL, Kapur V, Mehra R, Kuhlmann D, Fleishman SA, Ojile JM. Obstructive sleep apnea devices for out-of-center (OOC) testing: technology evaluation. J Clin Sleep Med. 2011 Oct 15;7(5):531-48. doi: 10.5664/JCSM.1328. PMID 22003351
- [Background] Aloia MS, Arnedt JT, Riggs RL, Hecht J, Borrelli B. Clinical management of poor adherence to CPAP: motivational enhancement. Behav Sleep Med. 2004;2(4):205-22. doi: 10.1207/s15402010bsm0204_3. PMID 15600056
- [Background] Chasens ER, Ratcliffe SJ, Weaver TE. Development of the FOSQ-10: a short version of the Functional Outcomes of Sleep Questionnaire. Sleep. 2009 Jul;32(7):915-9. doi: 10.1093/sleep/32.7.915. PMID 19639754
- [Background] Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. Circ Cardiovasc Qual Outcomes. 2015 Sep;8(5):469-76. doi: 10.1161/CIRCOUTCOMES.115.001958. PMID 26307129
- [Background] Aloia MS, Arnedt JT, Strand M, Millman RP, Borrelli B. Motivational enhancement to improve adherence to positive airway pressure in patients with obstructive sleep apnea: a randomized controlled trial. Sleep. 2013 Nov 1;36(11):1655-62. doi: 10.5665/sleep.3120. PMID 24179298
- [Background] Weaver TE , Crosby RD , Bron M , Menno D MS. Using Multiple Anchor-based And Distribution-based Estimates To Determine The Minimal Important Difference (MID) For The FOSQ-10. Sleep. 2018;41(Mid):292-293.
- [Background] WR, Miller, Rollnick S. Motivational Interviewing: Preparing People for Change. 2nd ed. New York: Guildford Press; 2002.
- [Background] Pena Orbea C, St Louis E, Dupuy-McCauley K, F Shaughnessy G, I Morgenthaler T. 0495 Sleep Medicine and the Hospitalized Patient: Evaluation and Predictors for Sleep Disordered Breathing Testing and Associated Outcomes. Vol 42.; 2019. doi:10.1093/sleep/zsz067.493